CLINICAL TRIAL: NCT03952728
Title: The Long-term Effects of an Intensive Lifestyle Intervention for Type 2 Diabetes on Medicare Eligibility, Health Care Use, and Health Care Spending
Brief Title: The Long-term Effects of an Intensive Lifestyle Intervention for Type 2 Diabetes on Medicare Outcomes
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of Southern California (Other); Wake Forest University (Other)
Responsible Party: Sponsor
Other Study IDs: UP-16-00706
Record Dates: First submitted 2018-12-13; First posted 2019-05-16 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ILI/ Treatment group: This group includes Look AHEAD participants who were initially assigned to the intensive lifestyle intervention, consented to administrative data linkages, and were successfully linked to Medicare databases.
  Interventions: Behavioral: Intensive lifestyle intervention
- Control group: This group includes Look AHEAD participants who were initially assigned to the diabetes support and education control arm, consented to administrative data linkages, and were successfully linked to Medicare databases.
  Interventions: Behavioral: Diabetes support and education

INTERVENTIONS:
Behavioral: Intensive lifestyle intervention — Lifestyle intervention focused on weight loss through diet and physical activity
  Groups: ILI/ Treatment group
Behavioral: Diabetes support and education — Behavioral intervention focused on diabetes support and education
  Groups: Control group

SUMMARY:
This study investigates whether an intensive lifestyle intervention for type 2 diabetes had long-term effects on Medicare enrollment, health care use, and health care spending.

DETAILED DESCRIPTION:
The Look AHEAD study tested whether participants with type 2 diabetes assigned to an intensive lifestyle intervention (ILI) for weight loss exhibited reductions in cardiovascular morbidity and mortality, relative to a control group receiving usual care and diabetes support and education. During the 12-year intervention period, the ILI led to persistent reductions in weight, waist circumference, and hemoglobin A1c and improvements in physical fitness. In addition, the ILI led to reductions in hospitalizations, hospital days, and prescription drug spending during the intervention period (through 2012). However, the longer-term effects (2012 and later) on health care use and spending remain unknown.

In an ongoing ancillary study, the researchers are investigating the effects of the ILI on economic outcomes, during and after the study. As a part of this study, the study team is linking consenting Look AHEAD participants to Medicare databases. The researchers will investigate the long-term effects of ILI on health care use and health care spending.

By 2012 nearly all Look AHEAD participants were eligible for Medicare due to age (over 65). To the extent that Look AHEAD participants developed severe disabilities, the participants may have gained Medicare eligibility earlier through enrollment in Social Security Disability Insurance (SSDI). Thus, the researchers will also test for differences in the Medicare enrollment channel between ILI and control group participants, specifically whether the groups enrolled through SSDI at different rates.

ELIGIBILITY:
Inclusion Criteria:

* Look AHEAD participation: met age requirements and other criteria at time of study enrollment (as noted in Look AHEAD Research Group (2013))
* Consented to administrative data linkages
* Provided individual identifiers that could be linked with Medicare databases
* Were successfully linked to Medicare data

Exclusion Criteria:

-

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes Look AHEAD participants that consented to administrative data linkages, provided individual identifiers that could be linked with Medicare data, and were successfully linked to Medicare data.
Sampling Method: Non-Probability Sample
Enrollment: 2796 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Total inpatient (general hospital/acute care) discharges | 12-years
  This is based on patient-level HEDIS specifications.
Total inpatient (general hospital/acute care) days | 12-years
  This is based on patient-level HEDIS specifications.
Total number of emergency department visits | 12-years
  This is based on patient-level HEDIS specifications.
Medicare Part D Prescription Drug Fill Count | 12-years
  Derived measure indicating number of 30-day supply equivalents in each year.

SECONDARY OUTCOMES:
Total Medicare spending | 12-years
  Sums Medicare payments across service use categories
Medicare inpatient payments | 12-years
  Patient-level inpatient payments
Medicare Part D drug payments | 12-years
  Part D plan payments for covered drugs in a given year
Medicare Part D drug costs | 12-years
  Gross drug costs for all Part D drugs for a given year
Medicare outpatient visits | 12-years
  Based on patient-level HEDIS specifications
Medicare hospital outpatient payments | 12-years
  Based on Medicare records
Medicare Part B physician payments | 12-years
  Based on Medicare records
Medicare Skilled Nursing Facility payments | 12-years
  Based on Medicare records

OTHER OUTCOMES:
Originally eligible for Medicare through Old Age and Survivor's Insurance | 12-years
  This is based on "Original Reason for Entitlement" field in Medicare Beneficiary Summary File
Originally eligible for Medicare through Disability Insurance Benefits | 12-years
  This is based on "Original Reason for Entitlement" field in Medicare Beneficiary Summary File
Originally eligible for Medicare due to End Stage Renal Disease (ESRD) | 12-years
  This is based on "Original Reason for Entitlement" field in Medicare Beneficiary Summary File
Hospital readmissions | 12-years
  Based on HEDIS specifications
Inpatient medicine discharges | 12-years
  Based on patient-level HEDIS specifications
Inpatient surgical discharges | 12-years
  Based on patient-level HEDIS specifications
Inpatient medicine days | 12-years
  Based on patient-level HEDIS specifications
Inpatient surgical days | 12-years
  Based on patient-level HEDIS specifications
Medicare Dialysis Payments | 12-years
  Based on Medicare records
Medicare Durable Medical Equipment payments | 12-years
  Based on Medicare records
Medicare Imaging + Test payments | 12-years
  Based on Medicare records

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Huckfeldt, PhD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: No
Use of Medicare data is restricted under a data use agreement between the Centers of Medicare and Medicaid Services and University of Southern California, Wake Forest, and the University of Minnesota.

REFERENCES:
- [Background] Look AHEAD Research Group; Wing RR, Bolin P, Brancati FL, Bray GA, Clark JM, Coday M, Crow RS, Curtis JM, Egan CM, Espeland MA, Evans M, Foreyt JP, Ghazarian S, Gregg EW, Harrison B, Hazuda HP, Hill JO, Horton ES, Hubbard VS, Jakicic JM, Jeffery RW, Johnson KC, Kahn SE, Kitabchi AE, Knowler WC, Lewis CE, Maschak-Carey BJ, Montez MG, Murillo A, Nathan DM, Patricio J, Peters A, Pi-Sunyer X, Pownall H, Reboussin D, Regensteiner JG, Rickman AD, Ryan DH, Safford M, Wadden TA, Wagenknecht LE, West DS, Williamson DF, Yanovski SZ. Cardiovascular effects of intensive lifestyle intervention in type 2 diabetes. N Engl J Med. 2013 Jul 11;369(2):145-54. doi: 10.1056/NEJMoa1212914. Epub 2013 Jun 24. PMID 23796131
- [Result] Huckfeldt PJ, Frenier C, Pajewski NM, Espeland M, Peters A, Casanova R, Pi-Sunyer X, Cheskin L, Goldman DP. Associations of Intensive Lifestyle Intervention in Type 2 Diabetes With Health Care Use, Spending, and Disability: An Ancillary Study of the Look AHEAD Study. JAMA Netw Open. 2020 Nov 2;3(11):e2025488. doi: 10.1001/jamanetworkopen.2020.25488. PMID 33231638